CLINICAL TRIAL: NCT02742610
Title: Brief Mindfulness Cessation Training With EMA for Post-hospital Depressed Smokers
Brief Title: Smoking Cessation Intervention for Smokers With Depression Receiving Outpatient Psychiatric Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fordham University (Other)
Collaborators: Albert Einstein College of Medicine (Other); University of Texas at Austin (Other); William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA037364-01A1 (NIH)
Record Dates: First submitted 2016-02-03; First posted 2016-04-19 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness with Contingency Management (Experimental): The intervention (MSI-CM) will involve two individual pre-quit in-person sessions and two post-quit phone counseling sessions, a series of brief mindfulness trainings that will be delivered via smartphone, that prompts participants to practice a mindfulness exercise five times a day while abstinent during the 2-week incentivized abstinence period (using CM) plus an additional 2 weeks (without CM) following the participant's target quit date. The MSI-CM participants will be asked to provide CO video via smartphone twice daily with monetary incentives provided (CM). Participants will receive monetary incentives contingent on each confirmed CO level (less than 7 ppm) for the CM period. We will use CM as an adjunct strategy to enhance the efficacy of mindfulness training.
  Interventions: Behavioral: Mindfulness with Contingency Management
- Active Control (Active Comparator): Participants assigned to the control group will receive two individual pre-quit in-person sessions and two post-quit phone counseling sessions, similar to the MSI-CM except for mindfulness introduction/discussion. Participants in the control group will receive the same monetary incentives on average as the participants in the MSI-CM for submitting CO videos, regardless of CO levels (non-abstinent contingent), during the 2-week post-TQD period. Each participant in the group (the non-contingent CO group) will be yoked to a single participant (selected randomly with stratification) in the MSI-CM. The yoked participant receives the same amount of monetary incentives as his or her matched participant in the contingent CO (MSI-CM) group.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Mindfulness with Contingency Management
  Arms: Mindfulness with Contingency Management
Behavioral: Active Control
  Arms: Active Control

SUMMARY:
This study aims to develop a Mindfulness Smartphone Intervention with Contingency Management (MSI-CM) for smoking cessation that can be readily available to depressed smokers receiving outpatient psychiatric treatment. This project is expected to result in the development of an effective intervention that will produce preliminary data showing increased short-term cessation success in depressed smokers receiving outpatient psychiatric treatment. It is anticipated that this smoking cessation intervention will have potential for broad reach to outpatient psychiatric treatment programs and have a significant overall impact in reducing smoking-related morbidity and mortality by enhancing smoking cessation rates in at-risk populations.

DETAILED DESCRIPTION:
The proposed study will develop a Mindfulness Smartphone Intervention with Contingency Management (MSI-CM) for smoking cessation that can be readily available to depressed smokers receiving outpatient psychiatric treatment. The intervention will involve a series of brief mindfulness training that will be delivered via smartphone, that prompts patients to practice a mindfulness exercise multiple times a day while abstinent: 1) 10-days prior to their target quit date and 2) during the 2-week incentivized abstinence period (using CM) plus an additional 2 weeks (without CM) following their target quit date. We will use CM as an adjunct strategy to enhance the efficacy of mindfulness training due to its utility in producing short-term abstinence, so as to provide opportunities to practice mindfulness without smoking in one's natural environment. We will accomplish this objective by pursuing the following specific aims (in 2 phases):

Phase 1: To develop the MSI-CM intervention intended to improve smoking cessation success among depressed smokers receiving outpatient psychiatric treatment.

1a. We will collaborate with TelASK, Inc. to develop a prototype of a smartphone intervention (MSI-CM).

1b. We will conduct preliminary pilot testing of MSI-CM, in an iterative fashion, with 10 smokers receiving outpatient psychiatric treatment for depression.

Phase 2: To conduct a preliminary, randomized controlled trial (RCT) with depressed 60 smokers receiving outpatient psychiatric treatment.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years of age
* be current daily smokers (i.e., at least 5 cigarettes for the past 6 months)
* English-speaking
* motivated to quit smoking (i.e., "intent to quit in the next 3 months")
* have a diagnosis of depressive or bipolar disorders
* engaged in outpatient psychiatric treatment (i.e., has been receiving outpatient psychiatric treatment for at least 3 months AND has received counseling from social worker at outpatient psychiatric treatment clinic at least 3 times in the past 3 months)

Exclusion Criteria:

* acute psychiatric symptomatology which precludes study participation including current active suicidal ideation
* diagnosis of psychotic disorders
* current diagnosis of dementia or cognitive impairment sufficient to impair provision of informed consent or study participation
* patient's inability to provide consent for study participation due to his/her inability to demonstrate an understanding of study procedures as contained in the statement of informed consent, after no more than two explanations
* current clinical diagnosis of intellectual development disorder or autistic disorder
* current (non-nicotine) substance use disorder with the exception of individuals holding 6 months of sobriety and/or receiving treatment including counseling and medications (i.e. methadone, suboxone)
* intention to quit smoking using pharmacotherapy other than transdermal nicotine patches
* pregnant, breastfeeding, or planning to become pregnant within 6 months
* significant history of cardiovascular disease (a standard contraindication for nicotine patch use),
* patient does not have a stable home address where the research team could reliably reach patient, or
* regular (3 or more times in the past month) use of other tobacco products (i.e., cigars, cigarillos, chewing tobacco) or marijuana

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Smoking Status | 2-week, 4-week, and 3-month post-target quit date assessment visit
  Self-reports of smoking status and verification via CO will be collected at 2-week, 4-week, and 3-month (cotinine level) post-target quit date assessment. The main outcome analyses are based upon 7-day point prevalence abstinence (PPA). As a secondary approach, we will use the timeline followback (TLFB) procedure for assessing the longitudinal course of smoking outcomes. Our approach permits us to follow the standard NCI and NHLBI guidelines for measurement. Biochemical Verification. Self-reported abstinence will be verified by carbon monoxide (CO) analysis of breath samples (6 ppm cutoff) for abstinence of 24 hours to one week for 3-month follow-up. Values above the cutoff will be considered indicative of smoking.

CONTACTS AND LOCATIONS:
Overall Officials: Haruka Minami, Ph.D., Principal Investigator — Fordham Univeristy
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Minami H, Nahvi S, Arnsten JH, Brinkman HR, Rivera-Mindt M, Wetter DW, Bloom EL, Price LH, Richman EK, Betzler TF, Stockmal C, Donnelly R, McClain LM, Kennedy KA, Vieira C, Fine M, McCarthy DE, Thomas JG, Hecht J, Brown RA. A pilot randomized controlled trial of smartphone-assisted mindfulness-based intervention with contingency management for smokers with mood disorders. Exp Clin Psychopharmacol. 2022 Oct;30(5):653-665. doi: 10.1037/pha0000506. Epub 2021 Jul 22. PMID 34291992